CLINICAL TRIAL: NCT04094909
Title: Efficacy and Safety of Rh-endostatin（Endostar）Combined With Platinum-based Doublet Chemotherapy and Pembrolizumab as First Line Therapy in Patients With Advanced or Metastatic Non-small-cell Lung Cancer
Brief Title: Rh-endostatin Combined With Chemotherapy and Pembrolizumab for Advanced NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, Zhou Chengzhi, Professor, Guangzhou Institute of Respiratory Disease
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CROC1902
Record Dates: First submitted 2019-09-17; First posted 2019-09-19 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Staging IV NSCLC
Keywords: rh-endostatin; Pembrolizumab; NSCLC; Chemotherapy
MeSH Terms: interventions — pembrolizumab; Carboplatin; Cisplatin; Pemetrexed; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rh-endostatin + chemotherapy+Pembrolizumab (Experimental): The subjects are 186, including Squamous and Non-Squamous NSCLC. Squamous NSCLC receives rh-endostatin at a dose of 15mg/m2 for 5 days and 200 mg of pembrolizumab at day 1 in each cycle, repeating every 3 weeks till to PD or unacceptable toxicities. all the patients with squamous NSCLC also receive carboplatin (5U/AUC) or cisplatin ( 75mg/m2) and [nab]-paclitaxel (100mg/m2) for the first 4 cycles. For non-squamous NSCLC, rh-endostatin at dose of 15mg/m2 for 5 days, 200 mg of pembrolizumab at day 1 and pemetrexed (500mg/m2,d1) are given in each cycle, repeating every 3 weeks till to PD or unacceptable toxicities. Non-squamous NSCLC also receive carboplatin (5U/AUC) or cisplatin ( 75mg/m2) and pemetrexed (500mg/m2,d1) for the first 4 cycles.
  Interventions: Drug: Rh-endostatin

INTERVENTIONS:
Drug: Rh-endostatin — Squamous NSCLC: Rh-endostatin+Pembrolizumab+carboplatin or cisplatin +[nab]-paclitaxel during the treatment. Rh-endostatin+Pembrolizumab during the maintenance period.
  Non-squamous NSCLC: Rh-endostatin+Pembrolizumab+carboplatin or cisplatin +pemetrexed during the treatment. Rh-endostatin+Pembrolizumab + pemetrexed during the maintenance period.
  Other Names: Pembrolizumab; carboplatin; cisplatin; pemetrexed; [nab]-paclitaxel

SUMMARY:
The aim of this study was to investigate that efficacy and safety of rh-endostatin（Endostar）combined with platinum-based doublet chemotherapy and Pembrolizumab as first line therapy in patients with advanced or metastatic non-small-cell lung cancer.

DETAILED DESCRIPTION:
The study design is a single arm. The subjects are 186, including Squamous and Non-Squamous NSCLC. Squamous NSCLC receives rh-endostatin at a dose of 15mg/m2 for 5 days and 200 mg of pembrolizumab at day 1 in each cycle, repeating every 3 weeks till to PD or unacceptable toxicities. all the patients with squamous NSCLC also receive carboplatin (5U/AUC) or cisplatin ( 75mg/m2) and [nab]-paclitaxel (100mg/m2) for the first 4 cycles. For non-squamous NSCLC, rh-endostatin at a dose of 15mg/m2 for 5 days, 200 mg of pembrolizumab at day 1 and pemetrexed (500mg/m2,d1) are given in each cycle, repeating every 3 weeks till to PD or unacceptable toxicities. Non-squamous NSCLC also receive carboplatin (5U/AUC) or cisplatin ( 75mg/m2) and pemetrexed (500mg/m2,d1) for the first 4 cycles. The radiographic evaluation will be taken place at baseline, 6 and 12 weeks after treatment and every 9 weeks thereafter based on Recist 1.1, till to PD or unacceptable toxicities. After that, survival follow-up is going on every 3 months till to the death. The safety evaluation is based on CTCAE 4.0. In addition to the above, the examination of ct DNA and PD-L1 for tumor sample and peripheral blood is taken at the baseline, and also examination of ct DNA and PD-L1 for peripheral blood at week 6 and 12 of treatment and at the time of PD.

Primary endpoint: .PFS Secondary endpoints:OS,ORR,DCR and safety

ELIGIBILITY:
Inclusion Criteria:

1. Sign informed consent.
2. Patients aged 18 to 75.
3. According to the TNM staging of lung cancer in the 8th edition of the International Association for Lung Cancer Research and the Joint Committee on Cancer Classification of the United States, NSCLC with local advanced or metastatic stage (stage III B, III C or IV) confirmed by histology or cytology can not be treated surgically and can not be accepted by radical concurrent radiotherapy and chemotherapy.
4. There must be at least one measurable lesion.
5. ECOG PS was 0-1.
6. NSCLC with driving gene was negative.
7. Patients who had not received systemic radiotherapy or chemotherapy before or who had relapsed more than 6 months after the end of adjuvant chemotherapy were followed up.
8. Patient's survival more than 3months.
9. The liver and kidney function is normal.

Exclusion Criteria:

1. The subjects had cancerous meningitis.
2. Patients with active central nervous system (CNS) metastasis should be excluded. If the patients with CNS metastasis can be adequately treated and the neurological symptoms of the subjects can be restored to baseline level at least two weeks before enrollment (except for residual signs or symptoms related to CNS treatment), who can be participated in the study. In addition, patients who do not use corticosteroids, or receive prednisone (or equivalent) at a steady or decreasing dose of less than 10 mg/day.
3. Patients with active, known or suspected autoimmune diseases were excluded. Patients with type I diabetes mellitus, hypothyroidism requiring hormone replacement therapy, skin disorders requiring no systemic treatment (e.g., vitiligo, psoriasis or alopecia), or who are not expected to reappear without external triggers may be included.
4. Within 14 days before admission, subjects requiring systemic corticosteroids (dose equivalent to > 10 mg prednisone/day) or other immunosuppressive drugs were included. Patients who used inhaled or topical corticosteroids, and those who received corticosteroid replacement therapy at doses equal to more than 10 mg of prednisone per day, could participate in the study if there were no active autoimmune diseases.
5. Hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus antibody (HCV Ab) are positive, indicating acute or chronic infection.
6. According to chest X-ray examination, sputum examination and clinical examination, active pulmonary tuberculosis (TB) infection was judged. Patients with a history of active pulmonary tuberculosis infection in the previous year should be excluded even if they have been treated; patients with a history of active pulmonary tuberculosis infection more than a year ago should also be excluded unless the course and type of antituberculosis treatment previously used are proved to be appropriate.
7. Previous serious heart disease patients include congestive heart failure, uncontrollable high-risk arrhythmia, unstable angina pectoris, myocardial infarction, severe valvular disease and intractable hypertension.
8. Pregnant or lactating patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2020-02-06 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
PFS | 6-10 months
  from the enrolment to PD or death

SECONDARY OUTCOMES:
OS | 14-18 months
  from the enrolment to death

CONTACTS AND LOCATIONS:
Overall Officials: Likun Chen, professor, Principal Investigator — Sun Yat-sen University
Locations (1):
- Zhou Chengzhi, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No